CLINICAL TRIAL: NCT07137871
Title: Phase 1 Clinical Trial of Avasopasem in Patients With Metastatic Hormone Receptor Positive Breast Cancer With Progression on a CDK 4/6 Inhibitor and Hormonal Therapy (CTMS# 24-0096)
Brief Title: Clinical Trial of Avasopasem in Patients With Metastatic Hormone Receptor Positive Breast Cancer With Progression on a CDK 4/6 Inhibitor and Hormonal Therapy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Kate Lathrop, Associate Professor, The University of Texas Health Science Center at San Antonio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTMS# 24-0096; STUDY00000816 (Other: University of Texas Health Science Center San Antonio)
Record Dates: First submitted 2025-08-15; First posted 2025-08-22 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Breast Cancer Metastatic
Keywords: Hormone receptor positive; HR+, HER2 negative metastatic breast cancer; Disease progression
MeSH Terms: conditions — Disease Progression | interventions — avasopasem manganese

STUDY DESIGN:
Intervention Model Description: This is a single institution, non-randomized, phase 1 clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Metastatic Hormone Receptor Positive Breast Cancer (Experimental): This study is investigating the addition of a novel agent, Avasopasem (or GC4419), in patients with hormonal receptor positive (HR+) metastatic breast cancer with progression while on treatment with a cyclin-dependent kinase 4 and 6 (CDK4/6) inhibitor and an aromatase inhibitor.
  Interventions: Drug: Avasopasem

INTERVENTIONS:
Drug: Avasopasem — Avasopasem has also been shown to exhibit both antitumor effects as well as minimal toxicity. Participants are currently taking a CDK 4/6 inhibitor and hormonal therapy
  Other Names: GC4419

SUMMARY:
This study aims to evaluate the safety of avasopasem in combination with CDK 4/6 inhibitor and hormonal therapy in women with metastatic hormone receptor positive breast cancer, and to see if the addition of avasopasem improves the effectiveness of a CDK 4/6 inhibitor and hormonal therapy.

DETAILED DESCRIPTION:
This is a phase 1 non-randomized clinical trial of Avasopasem in patients with metastatic hormone receptor positive breast cancer with progression on first line therapy consisting of a CDK 4/6 inhibitor and hormonal therapy to determine the efficacy and safety of the addition of Avasopasem in patients with metastatic HR+ breast cancer with progression after first line treatment with hormonal therapy (an AI or fulvestrant) and a CDK 4/6 inhibitor (ribociclib or abemaciclib). Each treatment cycle will be 28 days and tumor assessment by imaging with CT scans of the chest, abdomen and pelvis will be performed every two cycles.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of HR+, HER2 negative metastatic breast cancer.
* Estrogen receptor (ER) and/or progesterone receptor (PR) expression positivity is defined as at least 10% of tumor cells nuclei positive by immunohistochemistry in the sample on testing.
* HER2 negative: defined as IHC staining of 0 or 1+. If HER2 overexpression is equivocal by IHC, defined as 2+, the tumor must be non-gene amplified by FISH (ratio <2 and HER2 copy number <4).
* Progression on treatment with a CDK 4/6 inhibitor and hormonal therapy in the metastatic setting

  * The CDK 4/6 inhibitor must be ribociclib or abemaciclib. Patients on palbociclib are not eligible.
  * Patient may have been on palbociclib previously but must have been stable on ribociclib or abemaciclib for at least three months prior to enrolling. In this case, the switch from palbociclib to either ribociclib or abemaciclib must have been of toxicity management and not progression of disease.
  * Hormonal therapy is defined as an aromatase inhibitor (anastrozole, letrozole, exemestane) or fulvestrant.
  * Patients on tamoxifen are not eligible.
  * Both men and pre/perimenopausal women must be on ovarian suppression with a luteinizing hormone-releasing hormone (LHRH) agonist.
* Patients must have measurable disease based on RECIST 1.1 criteria.
* Females of child-bearing potential (FOCBP) who engage in intercourse must agree to use adequate contraception (e.g., hormonal or an intrauterine device [IUD] or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 3 weeks following completion of therapy.

NOTE: A FOCBP is any woman who meets the following criteria:

* Has not undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy
* Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)

  * FOCBP must have a negative serum pregnancy test within 7 days prior to registration.
  * Patients must be ≥ 18 years of age at the time of signing consent.
  * Patients must have an estimated life expectancy of at least 12 weeks.
  * Patients must exhibit an ECOG performance status of 0 or 1.
  * Patients must have adequate organ and bone marrow function as defined below:

    * Leukocytes (WBC) ≥ 3,000/mcL
    * Absolute neutrophil count (ANC) ≥ 1000/mcL
    * Hemoglobin (Hgb) ≥ 7 g/dL
    * Platelets (PLT) ≥ 100,000/mcL
    * Total bilirubin < 1.5 x Institutional upper limit of normal (ULN); ≤ 3.0 x ULN for patients with Gilbert's syndrome
    * AST (SGOT)/ALT (SGPT) < 3 x institutional ULN, or < 5 x ULN if liver metastasis present
    * Creatinine < 1.5 Institutional ULN
  * Patients with treated brain metastases are eligible if follow-up brain imaging at least 6 weeks after central nervous system (CNS)-directed therapy shows no evidence of progression.
  * Patients must have sufficient samples available to meet Menarini Silicon Biosystems (MSB) specimen requirements.
  * Patients with known history or current symptoms of cardiac disease, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.
  * Patients must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients who have any systemic therapy in the metastatic setting except hormonal therapy in combination with a CDK 4/6 inhibitor. Previously palliative targeted radiation therapy is allowed. Bone targeting agents such as bisphosphonates and rank ligand inhibitors for metastatic breast cancer to the bone is also allowed prior and during this trial.
* Patients with untreated new or progressive brain metastases or leptomeningeal disease
* Use of concomitant nitrates and PDE5 inhibitors.
* Use of potent CYP3A4 inhibitors or inducers and not able to discontinue two weeks prior to enrolling onto the trial.
* Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints. Note: Patients with HIV or infectious hepatitis must exhibit well controlled disease with stable treatment regimen (where applicable) that in the opinion of the treating physician should not preclude them from participating in the study.
* Patients who are currently pregnant or breast feeding.
* Patients with a history of another invasive malignancy within 2 years of registration with the exception of local squamous cell or basal cell carcinoma of the skin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-10-02 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Determine Safety and Tolerability of Treatment | Day 1 through Day 28 (each cycle is 28 days, up to 4 months
  Determine the safety and tolerability of Avasopasem in combination with a CDK 4/6 inhibitor and hormonal therapy. Each cycle of treatment will be 28 days. Toxicity will be assessed starting on the first day of each 28-day treatment cycle, using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0, and the incidence, nature, and severity of adverse events will be determined.All women who receive at least one dose of Avasopasem will be considered as evaluable for any toxicity and safety endpoints, as well as disease response. Patient reported outcome (PRO's) for adverse events (AE) will also be reported on day one of each cycle.

SECONDARY OUTCOMES:
Clinical Benefit Ratio (CBR) with addition of Avasopasem | Day 1 through Day 28 (each cycle is 28 days, up to 4 months
  Clinical benefit is defined as the percentage of patients with metastatic cancer who achieve as documented complete response, partial response, or stable disease following therapeutic intervention in this trial. A clinical benefit rate of 20% observed at 4 months (the time point for tumor assessment by Copy number alteration (CNA) and 18F-fluoroestradiol Positron Emission Tomography (FES-PET) will represent a clinically meaningful response rate with the addition of Avasopasem.

OTHER OUTCOMES:
Patient reported outcomes using European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire Core 30) and EORTC) QLQ-C-30 and EORTC QLC-BR23 a breast cancer-specific quality of life questionnaire | Day 1 through Day 28 (each cycle is 28 days, up to 4 months
  When the EORTC QLQ-C30 and QLQ-BR23 are used together, they are scored according to the EORTC QLQ-C30 scoring manual. Scores are linearly transformed to a 0-100 scale, with higher scores on functional scales indicating a higher level of functioning, and higher scores on symptom scales indicating a higher level of symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Kate Lathrop, MD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- Mays Cancer Center, UT Health San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided